CLINICAL TRIAL: NCT05374486
Title: PFI-RP: Smart Co-robot System for Cost-Effective Patient-Centered Robotic Rehabilitation
Brief Title: EEG Brain-Machine Interface Control of an Upper-Limb Robotic Exoskeleton for Robot-Assisted Rehabilitation After Stroke
Acronym: NeuroExo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Houston (Other)
Collaborators: TIRR Memorial Hermann (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jose L.Contreras-Vidal, Ph.D., Hugh Roy and Lillie Cranz Cullen Distinguished Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G0501521; HSC-MS-20-1287 (Other: University of Texas Health Science Center)
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Stroke; Hemiparesis
MeSH Terms: conditions — Stroke; Paresis | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- NeuroExo (Experimental): NeuroExo is a device which includes a robotic exoskeleton that you were in your affected arm to assist you with arm movements, a headset that you wear on your head to measure your brain activity and detect your intention to move, and a graphical user interface that allows you to initiate and stop neurotherapy, and track your motor performance.
  Interventions: Device: NeuroExo co-robot neurorehabilitation system

INTERVENTIONS:
Device: NeuroExo co-robot neurorehabilitation system — In this longitudinal study, adult subjects with hemiparesis due to chronic stroke will receive robotic-assisted upper-arm training through an EEG-based BMI control of robotic exoskeleton to study the changes in upper extremity motor function, cortical plasticity (using the EEG). After one screening visit, two baseline visits for EEG signal screens, six onsite training sessions will be provided with the NeuroExo system, followed by 60 home therapy sessions (2 sessions per day, 5 days per week for 6 weeks). If the participant have completed at least 50 sessions of neurotherapy at home, the participant will complete a set of measurements to assess function of the affected upper arm and brain activity within 3 days after the last session for post-assessment visit, and one-month post follow-up session. The total amount of time for this study is 16-20 weeks.
  Other Names: Brain-Machine Interface; Brain-Computer Interface; Neurorobotics; Rehabilitation Robotics

SUMMARY:
The goal of this study is to develop a clinically feasible, low-cost, nonsurgical neurorobotic system for restoring function to motor-impaired stroke survivors that can be used at the clinic or at home. Moreover, another goal is to understand how physical rehabilitation assisted by robotic device combined with electroencephalograph (EEG) can benefit adults who have had stroke to improve functions of their weaker arm.

The proposed smart co-robot training system (NeuroExo) is based on a physical upper-limb robotic exoskeleton commanded by a non-invasive brain machine interface (BMI) based on scalp EEG to actively include the participant in the control loop .

The study will demonstrate that the Neuroexo smart co-robot arm training system is feasible and effective in improving arm motor functions in the stroke population for their use at home.The NeuroExo study holds the promise to be cost-effective patient-centered neurorehabilitation system for improving arm functions after stroke.

DETAILED DESCRIPTION:
This study has two phases: The first phase will consist of baseline recordings for system calibration and training sessions to be conducted in a clinical setting. The second phase will consist of NeuroExo BMI-exo neurotherapy to be conducted at the participant's home. Throughout the study and after completion of the study, movement and brain activity will be analyzed to assess function of the affected upper extremity and changes in brain activity associated with the neurotherapy.

ELIGIBILITY:
Inclusion Criteria:

* subjects between the ages of 20-65, male or female,
* mild-to- moderate unilateral stroke confirmed by brain CT or MRI scan and manifested by a Glasgow Coma scale (GCS) score between 15 and 9 documented within 6 months,
* the ability to perform 20deg of active wrist/elbow for upper limb robotic movement on the affected side, no planned alteration in lower/upper- extremity therapy/medication for muscle tone during course of study,
* Anticipated length of needed acute interdisciplinary rehabilitation of 30 days or more.
* Patients are required to have a MMSE>=24 to rule out those with cognitive impairments.
* Patients will have to have normal/near normal strength in one upper/lower extremity and appreciable weakness in the other upper/lower extremity.

Exclusion Criteria:

* history of traumatic brain injury prior to the current episode,
* Severe neurologic or psychiatric condition preventing participation in rehabilitation and physical therapy activities (patients unable or unwilling to receive instruction and effectively complete a simple assigned task as determined by MMSE>=24 specified in inclusion criteria).
* Women and minorities will be recruited as long as they meet the inclusion criteria.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Fugl-Meyer Arm (FMA) Motor Score | Baseline, immediately after end of treatment (within a week), and 4 weeks after end of treatment
  FMA is a stroke-specific, performance based impairment index. It quantitatively measures impairment based on Twitchell and Brunnstrom's concept of sequential stages of motor return in hemiplegic stroke patients. It uses an ordinal scale for scoring of 33 items for the upper limb component of the F-M scale (0:can not perform; 1:can perform partially; 2:can perform fully). Total range is 0-66, 0 being poor and 66 normal.
Neural Activity (Cortical Dynamics) Measured by Electroencephalography (EEG) Movement-related Cortical Potential (MRCP) Amplitude | Baseline, immediately after end of treatment (within a week), and 4 weeks after end of treatment
  EEG activity in the delta, theta, alpha, beta and gamma bands will be assessed. Scalp EEG electrodes will be located over the motor cortex, specifically, central (Cz, C1- C4), fronto- central (FCz, FC1 - FC4) and centro-parietal electrodes (CPz, CP1 - CP4). Further, to account for left hand vs. right hand impairment, the electrode locations will be flipped for individuals with right hand impairment. Increased MRCP amplitude indicates increased activation of the ipsi-lesional hemisphere or inhibition of competing contra-lesional hemisphere, following motor relearning.
Cortical Dynamics Measured by Electroencephalography (EEG) Movement-related Cortical Potential (MRCP) Latency | Baseline, immediately after end of treatment (within a week), and 4 weeks after end of treatment
  EEG activity in the low-frequency delta band will be assessed. Scalp EEG electrodes will be located over the motor cortex, specifically, central (Cz, C1- C4), fronto- central (FCz, FC1 - FC4) and centro-parietal electrodes (CPz, CP1 - CP4). Further, to account for left hand vs. right hand impairment, the electrode locations will be flipped for individuals with right hand impairment. MRCP latency is the duration of MRCP prior to movement onset, and is defined as time difference starting from 50% of peak amplitude until the time of movement onset. Increased MRCP latency indicates increased activation of the ipsi-lesional hemisphere or inhibition of competing contra-lesional hemisphere, following motor relearning.
Movement Quality as Assessed by Exoskeleton Kinematics | Baseline, immediately after end of treatment (within a week), and 4 weeks after end of treatment
  A higher value indicates better movement quality.
Movement Quality as Assessed by Exoskeleton Kinematics - Number of Peaks | Baseline, immediately after end of treatment (within a week), and 4 weeks after end of treatment
  Number of peaks is a metric related to the shape of the velocity profile. A higher number of peaks implies jerkier movement. A lower number of peaks indicates better movement quality (that is, movements are less jerky).
Movement Quality as Assessed by Exoskeleton Kinematics - Time to First Peak | Baseline, immediately after end of treatment (within a week), and 4 weeks after end of treatment
  Time to 1st Peak is a metric related to the shape of the velocity profile, and is reported as [(time to first peak) divided by (total movement duration)]. This value is usually less than the ideal value of 0.5, or 50%, of the total movement duration when a movement has more than one peak. The closer the value is to the ideal value of 0.5, the more well-balanced are the movements.

SECONDARY OUTCOMES:
Score on Action Research Arm Test (ARAT) | Baseline, immediately after end of treatment (within a week), and 4 weeks after end of treatment
  The ARAT is used to assess subject's ability to manipulate-lift-release objects horizontally and vertically, which differs in size, weight and shape. The test consists of 19 items divided into 4 sub-tests (grasp, grip, pinch, gross arm movement) and each item is rated on a 4-point scale. The possible total score ranges between 0-57. Higher scores indicate better performance.
Score on Jebsen-Taylor Hand Function Test (JTHFT) | Baseline, immediately after end of treatment (within a week), and 4 weeks after end of treatment
  The JTHFT is a motor performance test and assesses the time needed to perform 7 everyday activities (for example, flipping cards and feeding). Score is reported as items completed per second.
Grip Strength | Baseline, immediately after end of treatment (within a week), and 4 weeks after end of treatment
  A grip dynamometer will be used to measure maximum gross grasp force.
Pinch Strength | Baseline, immediately after end of treatment (within a week), and 4 weeks after end of treatment
  A pinch gauge will be used to measure maximum pinch force.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Contreras-Vidal, PhD, Principal Investigator — University of Houston; Gerard Francisco, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (3):
- United States (3):
  - The Institute for Rehabilitation and Research (TIRR) at Memorial Hermann, Houston, Texas
  - TIRR Memorial Hermann Hospital, Houston, Texas
  - University of Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Background] Bhagat NA, Yozbatiran N, Sullivan JL, Paranjape R, Losey C, Hernandez Z, Keser Z, Grossman R, Francisco GE, O'Malley MK, Contreras-Vidal JL. Neural activity modulations and motor recovery following brain-exoskeleton interface mediated stroke rehabilitation. Neuroimage Clin. 2020;28:102502. doi: 10.1016/j.nicl.2020.102502. Epub 2020 Nov 19. PMID 33395991
- [Background] Sullivan JL, Bhagat NA, Yozbatiran N, Paranjape R, Losey CG, Grossman RG, Contreras-Vidal JL, Francisco GE, O'Malley MK. Improving robotic stroke rehabilitation by incorporating neural intent detection: Preliminary results from a clinical trial. IEEE Int Conf Rehabil Robot. 2017 Jul;2017:122-127. doi: 10.1109/ICORR.2017.8009233. PMID 28813805
- [Background] Bhagat NA, Venkatakrishnan A, Abibullaev B, Artz EJ, Yozbatiran N, Blank AA, French J, Karmonik C, Grossman RG, O'Malley MK, Francisco GE, Contreras-Vidal JL. Design and Optimization of an EEG-Based Brain Machine Interface (BMI) to an Upper-Limb Exoskeleton for Stroke Survivors. Front Neurosci. 2016 Mar 31;10:122. doi: 10.3389/fnins.2016.00122. eCollection 2016. PMID 27065787
- [Background] Bhagat NA, French J, Venkatakrishnan A, Yozbatiran N, Francisco GE, O'Malley MK, Contreras-Vidal JL. Detecting movement intent from scalp EEG in a novel upper limb robotic rehabilitation system for stroke. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:4127-4130. doi: 10.1109/EMBC.2014.6944532. PMID 25570900
- [Background] Venkatakrishnan A, Francisco GE, Contreras-Vidal JL. Applications of Brain-Machine Interface Systems in Stroke Recovery and Rehabilitation. Curr Phys Med Rehabil Rep. 2014 Jun 1;2(2):93-105. doi: 10.1007/s40141-014-0051-4. PMID 25110624